CLINICAL TRIAL: NCT05593679
Title: A Multi-center Registry for Clinical Information and 99mTc-pyrophosphate Scintigraphy in Patients With Suspected Cardiac Amyloidosis in Taiwan
Brief Title: A Multi-center Cardiac PYP Scan Registry in Taiwan
Status: Recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 111229-E
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Cardiac Amyloidosis
MeSH Terms: conditions — Heart Failure; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tc-99m PYP Cardiac scan — Tc-99m PYP Cardiac scan

SUMMARY:
Amyloid deposition in the heart is called cardiac amyloidosis (CA); 95% is immunoglobulin light chain amyloidosis (AL) and transthyretin amyloidosis (ATTR). Hereditary (ATTRm) or wild-type (ATTRwt) depends on whether the ATTRm gene is mutated or not. The most common mutation in Taiwan is A97S, 80% have left ventricular hypertrophy. The good prognosis depends on early diagnosis and correct treatment strategy.

Bone-avid tracers such as 99mTc-PYP/DPD/HMDP could detect CA. The mechanism is not clear yet, which may be related to the microcalcification. AL amyloidosis is mostly between visual score grade 0-2, and ATTR-CM is usually grade≥2 on PYP scan, or heart to contralateral (H/CL) ratio, and it might replace invasive myocardial biopsy. However, there are no large-scale clinical studies, lack of standardization data, and limited information in comparison between clinical and imaging parameters.

The project will enroll patients with suspected or diagnosed with CA according to CA diagnostic algorithm. Clinical data and image parameters are collected and compared. The project aims to set up prediction models based on the multi-parameters of PYP scan using artificial intelligence technology, including imaging registration and alignment technology, and standardization. The investigators further use the key cardiovascular data elements and imaging-derived database using model training network to extract image features to develop the diagnostic and prognostic prediction models, which are expected to validate the clinical significance and improve patient-centric performance and efficient clinical decision making.

DETAILED DESCRIPTION:
The investigators will retrospectively and prospectively collect total PYP scans that had been performed on suspected or diagnosed ATTR-CM patients in medical centers in Taiwan and follow-up at least 1 year. You are enrolled based on clinical suspicions such as "red-flag" signs using ultrasound, NT-pro BNP and clinical data according to the diagnostic algorithms. If you are with Grade 2 and 3 PYP myocardial uptake, genetic testing is arranged, serum and urine AL tests results will be confirmed. Before reading, the imaging quality will be evaluated (good quality, fair but interpretable, poor but interpretable, poor and insufficient for interpretation). All the images will be visually graded by experienced nuclear medicine physicians with consensus. It helps understand the real-world data.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 20 years of age
2. Documented diagnosis or r/o of ATTR amyloidosis

Exclusion Criteria:

1. Pregnant or nursing (lactating) women.
2. Important systemic diseases (except heart disease or neurological diseases) such as liver cirrhosis, active malignant tumors, etc., with a life expectancy of less than 6 months.
3. Patient who refused clinical follow up.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients screened for ATTR-CM
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-08-29 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | 1 year
  Death

SECONDARY OUTCOMES:
CV death | 1 year
  CV death
Hospitalization for heart failure | 1 year
  Hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Wen Wu, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-31): https://cdn.clinicaltrials.gov/large-docs/79/NCT05593679/Prot_SAP_000.pdf